CLINICAL TRIAL: NCT00425802
Title: A Non-Myeloablative Conditioning Regimen With Peri-Transplant Rituximab and the Transplantation of Hematopoietic Stem Cells From HLA-Compatible Related or Unrelated Donors in Patients With B Cell Lymphoid Malignancies
Brief Title: Chemotherapy, Total-Body Irradiation, Rituximab, and Donor Stem Cell Transplant in Treating Patients With B-Cell Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-150; MSKCC-06150
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-02

CONDITIONS: Leukemia; Lymphoma
Keywords: noncontiguous stage II adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large-Cell, Immunoblastic | interventions — Antilymphocyte Serum; Filgrastim; Rituximab; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Whole-Body Irradiation

ARMS (1):
- treatment (Other): This is a phase 2 study of a treatment regimen consisting of a non-myeloablative (NMA) conditioning regimen incorporating low dose chemotherapy and low dose radiation as well as peri-transplant Rituximab and the transplantation of peripheral blood stem cells (PBSC) or bone marrow if PBSC collection not possible from an HLA compatible related or unrelated donor in patients with B cell lymphoid malignancies including diffuse large cell (DLC) and mantle cell non-Hodgkin's lymphoma (NHL), indolent B cell NHL, or chronic lymphocytic leukemia (CLL).
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Biological: graft-versus-tumor induction therapy; Biological: rituximab; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Biological: graft-versus-tumor induction therapy
Biological: rituximab
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. Also, monoclonal antibodies, such as rituximab, can find cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving rituximab before transplant and cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase II trial is studying the side effects and how well giving chemotherapy and radiation therapy together with rituximab and donor stem cell transplant works in treating patients with B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * CD20-positive aggressive B-cell non-Hodgkin's lymphoma (NHL), including any of the following subtypes:

    * Diffuse large cell lymphoma*, meeting 1 of the following criteria:

      * Relapsed disease after initial therapy, but failed to mobilize or had bone marrow involvement and therefore is not suitable for an autologous stem cell transplantation
      * High-intermediate- or high-risk second-line, age-adjusted International Prognostic Index score and in second complete remission (CR) or partial remission (PR) after autologous stem cell transplantation
      * Failed prior autologous stem cell transplantation and in PR or better after salvage chemotherapy
    * Large cell transformation of indolent NHL or chronic lymphocytic leukemia (CLL), meeting the following criteria:

      * In CR or PR of the large cell component of disease after salvage chemotherapy or autologous stem cell transplantation
    * Mantle cell lymphoma*, meeting 1 of the following criteria:

      * High-risk disease (e.g., p53 positivity) and in first CR or PR after initial therapy
      * Relapsed disease after initial therapy and in second or third CR or PR after salvage chemotherapy NOTE: *No progressive disease at allograft work-up
  * CD20-positive indolent NHL (e.g., follicular lymphoma, small cell lymphoma, or marginal zone NHL) OR CLL

    * Second or subsequent progression (pre-allograft cytoreduction necessary, but CR or PR not required)
* Relapsed disease must be biopsy-proven
* Must have received pre-allograft salvage chemotherapy, including 1 of the following:

  * Single autologous stem cell transplantation using high-dose chemotherapy conditioning within the past 120 days
  * At least 2 courses of intensive combination chemotherapy (e.g., RICE [rituximab, ifosfamide, carboplatin, etoposide]), according to diagnosis, within the past 80 days
  * CLL patients who have received CAMPATH do not have to receive pre-allograft salvage chemotherapy
* HLA-compatible related or unrelated donor available

  * HLA-matched ≥ 9/10 of the A, B, C, DRB1, and DQB1 loci, as tested by high resolution typing

    * One allele mismatch allowed

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Creatinine < 1.2 mg/mL OR creatinine clearance ≥ 50 mL/min
* Bilirubin < 2.5 mg/dL
* AST and ALT ≤ 3 times upper limit of normal (unless benign congenital hyperbilirubinemia is present)
* Spirometry and corrected DLCO ≥ 50% of normal
* LVEF ≥ 40%
* Albumin ≥ 2.5 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active uncontrolled infection, including active infection with Aspergillus or other mold
* No HIV infection
* No hepatitis B antibody or antigen positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior allogeneic transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-11-28 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo R. Castro-Malaspina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Juliet Barker, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center; Craig Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Sauter CS, Lechner L, Scordo M, Zheng J, Devlin SM, Fleming SE, Castro-Malaspina H, Moskowitz CH. Pretransplantation fluorine-18-deoxyglucose--positron emission tomography scan lacks prognostic value in chemosensitive B cell non-hodgkin lymphoma patients undergoing nonmyeloablative allogeneic stem cell transplantation. Biol Blood Marrow Transplant. 2014 Jun;20(6):881-4. doi: 10.1016/j.bbmt.2014.02.009. Epub 2014 Feb 15. PMID 24534109
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 11/28/2006 Protocol Closed to Accrual 4/22/2014 Primary Completion Date 10/28/2016 Recruitment Location is the medical clinic
Period: Overall Study
Arm/Group | Treatment
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 61
Age, Continuous [Median (Full Range); unit: years] | 54 [33 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 59
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 1 Year
Time Frame: 1 year
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 51
percentage of participants | 90 [81 to 98]

2. Secondary Outcome: Time to Neutrophil Engraftment
Time Frame: 2 years
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Median (Full Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 51
days | 15 [10 to 25]

3. Secondary Outcome: Time to Platelet Engraftment
Time Frame: 1 year
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Median (Full Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 51
days | 12 [6 to 40]

4. Secondary Outcome: Incidence of Moderate to Severe Grades II to IV Graft Versus Host Disease (GVHD) at 100 Days
Time Frame: 100 days
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 51
percentage of patients | 18 [7 to 29]

5. Secondary Outcome: Incidence of Chronic GVHD at 1 Year
Time Frame: 1 year
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 51
percentage of participants | 14 [3 to 24]

6. Secondary Outcome: Immune Reconstruction/CD4+ Count at 3 Months
Time Frame: 3 months
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Median (Inter-Quartile Range); unit: cells/microliters
Arm/Group | Treatment
Number analyzed (Participants) | 51
cells/microliters | 253 [160 to 343]

7. Secondary Outcome: Response to Treatment
Time Frame: 2 years
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 51
Participants
  Complete Response | 22
  Partial Response | 17
  Stable Disease | 11
  Progression of Disease | 1

8. Secondary Outcome: Immune Reconstruction/CD4+ Count at 6 Months
Time Frame: 6 months
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Median (Inter-Quartile Range); unit: cells/microliter
Arm/Group | Treatment
Number analyzed (Participants) | 51
cells/microliter | 312 [174 to 457]

9. Secondary Outcome: Immune Reconstruction/CD4+ Count at 1 Year
Time Frame: 1 year
Population: Data for the remaining 10 patients was not fully collected or analyzed for publication
Measure: Median (Inter-Quartile Range); unit: cells/microliter
Arm/Group | Treatment
Number analyzed (Participants) | 51
cells/microliter | 333 [18 to 1317]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 9/61
Serious Adverse Events (participants affected / at risk) | 26/61
Other Adverse Events (participants affected / at risk) | 59/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=61)
Hyperbilirubinemia (Investigations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Confusion (Psychiatric disorders) | 1
Death Not Otherwise Specified (General disorders) | 1
Death not assoc w CTCAE term - Disease progression (General disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Gait disturbance (General disorders) | 1
Fatigue (General disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Fever (in the absence of neutropenia) (General disorders) | 8
Gastrointestinal, other (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Infection - catheter related (Infections and infestations) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Infection, other (Infections and infestations) | 7
Mucositis - oral (Gastrointestinal disorders) | 1
Neurology - other (Nervous system disorders) | 1
Sensory neuropathy (Nervous system disorders) | 1
Ocular/visual - other (Eye disorders) | 1
Ophthalmoplegia/Diplopia (double vision) (Eye disorders) | 1
Lymphocytopenia (Investigations) | 1
Headache (Nervous system disorders) | 1
Pain - oral cavity (Gastrointestinal disorders) | 1
Phlebitis (Vascular disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Renal failure (Renal and urinary disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
Chills (General disorders) | 1
Seizure (Nervous system disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=61)
Infection, other (Infections and infestations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 26
Creatinine (Investigations) | 25
Alanine Aminotransferase (Investigations) | 13
Aspartate Aminotransferase (Investigations) | 13
Bilirubin (Investigations) | 7
Alkaline phosphatase (Investigations) | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes